CLINICAL TRIAL: NCT00390650
Title: An Eight-Week, Multicenter, Randomized, Double-blind, Placebo-controlled Study, With Escitalopram as an Active Control, to Evaluate the Efficacy, Safety and Tolerability of a Saredutant 100 mg Dose Once Daily, in Patients With Generalized Anxiety Disorder
Brief Title: A North-American Eight-week Study to Evaluate the Efficacy and Safety of Saredutant in Patients With Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5581; SR48968
Record Dates: First submitted 2006-10-19; First posted 2006-10-20 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-04

CONDITIONS: Anxiety
Keywords: Anxiety; clinical trials
MeSH Terms: conditions — Anxiety Disorders | interventions — SR 48968

INTERVENTIONS:
Drug: Saredutant

SUMMARY:
The primary objective is to evaluate the efficacy of a 100 mg dose of saredutant compared to placebo in patients with generalized anxiety disorder. The secondary objectives are to evaluate the efficacy of saredutant on disability and quality of life in patients with generalized anxiety disorder, and to evaluate blood levels of saredutant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of generalized anxiety disorder as defined by Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) criteria and confirmed by the Mini International Neuropsychiatric Interview (MINI) Plus Generalized Anxiety Disorder module.

Exclusion Criteria:

* Total score of less than 22 on the HAM-A.
* Montgomery-Asberg Depression Rating Scale (MADRS) total score greater than 18.
* Patients with a current history (within 6 months) of major depressive disorder or history or presence of bipolar disorders or psychotic disorders.
* Patients with alcohol dependence or abuse or substance dependence or abuse in the past 12 months except nicotine or caffeine dependence.
* Patients who have used the following prior to entry into Acute Phase: antipsychotics within 3 months, antidepressants including Monoamine Oxidase Inhibitors (MAOIs) within 1 month, anxiolytics within 2 weeks, mood-stabilizer (lithium, anticonvulsants) within 1 month, and/or high dose or prolonged benzodiazepine (continuous use for 3 months prior to admission) use.

The investigator will evaluate whether there are other reasons why a patient may not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2006-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study is the change from baseline to Day 56 of treatment in the Hamilton Anxiety Rating Scale (HAM-A) total score.

SECONDARY OUTCOMES:
The key secondary efficacy outcome is change from baseline in the Clinical Global Impression Severity of Illness score.

CONTACTS AND LOCATIONS:
Overall Officials: Marie TRAD, MD, Study Director — Sanofi
Locations (2):
- Sanofi-Aventis, Bridgewater, New Jersey, United States
- Sanofi-Aventis, Laval, Canada

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com